CLINICAL TRIAL: NCT04755010
Title: "De Novo" Atrial Fibrillation in Patients With Heart Failure: Incidence; Predictors and Relevance.
Acronym: FAISCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: University of Salamanca (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Principal Investigator, Moises Rodriguez Mañero, MD,PhD, Hospital Clinico Universitario de Santiago
Other Study IDs: 2019/082
Record Dates: First submitted 2020-11-11; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Implantable cardiac monitoring
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological characterization
  Human plasma samples: Total venous blood samples (10 ml) will be collected in EDTA tubes as anticoagulant and separated by centrifugation at 1500xg during 15 minutes plasma and cellular fractions. The supernatant and the cell pellet are transferred to tubes and stored at -80°C. The serological samples will be stored in each center of origin. Several determinations will be performed:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Linq II implantable cardiac monitor — Implantation of Linq II implantable cardiac monitor

SUMMARY:
Atrial fibrillation (AF) represents a problem of great implications to patients with heart failure (HF). Therefore, the risk of having AF increases up to 4,5 -5,9 times with the presence of HF. Both conditions share risk factors and the presence of the one worsens the progress of the other. Therefore, the AF is not only relevant in terms of thromboembolic events. Timing of AF progression seems to be associated with an increase in all causes of mortality. Although, it is estimated that between 30%-40% of the patients with HF develop AF, given that in many cases it occurs with no apparent symptoms for the patients, is considered that the number of affected patients is greater. Since silent AF poses a problem of great impact in patients with HF, monitoring through continuous electrocardiographic registry could be useful in those patients with a higher risk of thromboembolic events. The purpose of this study is to understand the mechanism and biological and clinical relevance of the AF from a holistic approach. Trying to distinguish the symptomatic AF from the silent one using the implementation of insertable cardiac devices. The purpose of this study is 1. To determine in which percentage of patients with HF, episodes of AF both symptomatic and asymptomatic occur, as well as if the presence of AF represents an irrelevant fact in the progression of the insufficiency or in the contrary, it is the cause of the HF patients clinical decline. 2. To examine the presence of triggers of AF in patients with HF and to identify the presence of clinical markers, image markers of the atrium and left ventricle, as well as biomarkers which allow the risk of stratification and could mean future therapeutic targets.

DETAILED DESCRIPTION:
Multicenter prospective study formed by units with experience in the management of patients with HF (Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Spain; Hospital Clínico Universitario de Salamanca, Salamanca, Spain and Hospital Universitario Virgen de la Arrixaca, Murcia, Spain).

Based on an AF development estimate of 30%, it has been estimated a minimum follow-up of 18 months and a maximum of 36 months for obtaining robust conclusions. On the basis of previously reported data, it has been estimated that the annual rate of AF in patients 65 years of age or older who have CHA2DS2VASc ≥ 2 and who have received an ICM is 6%. The enrolment of 300 patients had been estimated. The study would have 95% power to detect an episode of rapid atrial rate.

Those patients with a CHA2DS2VASc ≥2 seen in the HF unit will be prospectively included. In these patients, the previous diagnosis of AF will be assessed by means of clinical history and medical records. Patients with previous AF will be excluded.

Patients with preserved or intermediate LVEF will be defined according to current guidelines.

* Patients with signs and symptoms of HF.
* LVEF between 40 and 49 for "mid-range" and greater than or equal to 50 for those with LVEF preserved and at least one of these two criteria:

  * High natriuretic peptides (BNP> 35 pg / ml and / or NT-proBNP> 125 pg / mL)
  * Relevant structural disease (left ventricular hypertrophy or dilatation left earphone).
  * Diastolic dysfunction.

The data will be collected individually by each recruiting center and introduced in the online registration form that will be enabled (see next point). The definition of variables will be agreed upon among all recruiting centers. The information collected will be dumped into a database created specifically for this purpose and will be coordinated from the Hospital Clínico de Santiago de Compostela.

Remote monitoring The CareLink remote monitoring system allows remote monitoring of patients, without the need to go to the hospital center. This system establishes a connection between the patient and the medical center, through the patient monitor that reads the information from the implanted device and transmits it to a secure server. This communication allows the transmission of clinically significant events or, in the case of wireless devices, the sending of alerts. In this way, the healthcare professional has information of the event and allows him to anticipate the evaluation and treatment with the consequent benefit for the patient.

Biological characterization

Human plasma samples: Total venous blood samples (10 ml) will be collected in EDTA tubes as anticoagulants and separated by centrifugation at 1500xg during 15 minutes plasma and cellular fractions. The supernatant and the cell pellet are transferred to tubes and stored at -80°C. The serological samples will be stored in each center of origin. Several determinations will be performed:

ELIGIBILITY:
Inclusion Criteria:

* Patients with the previous diagnosis of HF with both preserved and depressed LVEF. Patients with preserved or intermediate LVEF will be defined according to current guidelines.

  1. Patients with signs and symptoms of HFor b) LVEF between 40 and 49 for "mid range" and greater than or equal to 50 for those with LVEF preserved, high natriuretic peptides (BNP> 35 pg / ml and / or NT-proBNP> 125 pg / mL)and at least one of these two criteria: Relevant structural disease (left ventricular hypertrophy or dilatation left earphone).

Diastolic dysfunction.

Exclusion Criteria:

* Previous history of atrial fibrillation.
* CHA2DS2VASc < 2.
* Patients requiring ventricular pacing > 40 patients
* Patients under cardiac resynchronization therapy pacemaker/devices.
* Patients with severe valvulopathy.
* Patients with reverseble

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: On the basis of previously reported data, we estimated that the annual rate of AF in patients 65 years of age or older who have CHA2DS2VASc ≥ 2 and who have received an ICM or a pacemaker would be approximately 6%. We then estimated that with enrolment of 300 patients, the study would have 95% power to detect an episode of rapid atrial rate
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AF | 3 years
  Prevalence and predictor of atrial fibrillation in 300 patients with heart failure and without previous history of AF determined by the Reveal LINQ Insertable Cardiac Monitor

SECONDARY OUTCOMES:
Echocardiography | 3 years
  Number of patients with heart failure with low late left atrial strain rate and atrial fibrillation versus patients with normal left atrial strain determined by the Reveal LINQ Insertable Cardiac Monitor

CONTACTS AND LOCATIONS:
Overall Officials: moises rodriguez mañero, PhD, Principal Investigator — Clínico Universitario de Santiago de Compostela
Locations (1):
- Moises Rodriguez Mañero, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data will be collected individually by each recruiting center and introduced in the online registration form that will be enabled.
  Information collection will be dumped into a database created specifically for this purpose and will be coordinated from the Hospital Clínico de Santiago de Compostela.

REFERENCES:
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Background] Healey JS, Alings M, Ha A, Leong-Sit P, Birnie DH, de Graaf JJ, Freericks M, Verma A, Wang J, Leong D, Dokainish H, Philippon F, Barake W, McIntyre WF, Simek K, Hill MD, Mehta SR, Carlson M, Smeele F, Pandey AS, Connolly SJ; ASSERT-II Investigators. Subclinical Atrial Fibrillation in Older Patients. Circulation. 2017 Oct 3;136(14):1276-1283. doi: 10.1161/CIRCULATIONAHA.117.028845. Epub 2017 Aug 4. PMID 28778946
- [Background] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Wachter R, Pouliot E, Ziegler PD; REVEAL AF Investigators. Incidence of Previously Undiagnosed Atrial Fibrillation Using Insertable Cardiac Monitors in a High-Risk Population: The REVEAL AF Study. JAMA Cardiol. 2017 Oct 1;2(10):1120-1127. doi: 10.1001/jamacardio.2017.3180. PMID 28842973
- [Background] Piccini JP, Passman R, Turakhia M, Connolly AT, Nabutovsky Y, Varma N. Atrial fibrillation burden, progression, and the risk of death: a case-crossover analysis in patients with cardiac implantable electronic devices. Europace. 2019 Mar 1;21(3):404-413. doi: 10.1093/europace/euy222. PMID 30462208
- [Background] DeCicco AE, Finkel JB, Greenspon AJ, Frisch DR. Clinical significance of atrial fibrillation detected by cardiac implantable electronic devices. Heart Rhythm. 2014 Apr;11(4):719-24. doi: 10.1016/j.hrthm.2014.01.001. Epub 2014 Jan 3. PMID 24394157